CLINICAL TRIAL: NCT00447356
Title: Phase III Randomized Study of Four Weeks High Dose IFN-2b in StageT3-T4 or N1 (Microscopic) Melanoma
Brief Title: High-Dose Interferon Alfa in Treating Patients With Stage II or StageIII Melanoma
Status: Withdrawn | Phase: Phase 3 | Type: Interventional
Why Stopped: There were no patient enrolled in this study at this site
Sponsor: Hackensack Meridian Health (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: E1697
Record Dates: First submitted 2007-03-12; First posted 2007-03-14 (Estimated); Last update posted 2013-05-13 (Estimated); Status verified 2013-05

CONDITIONS: Melanoma (Skin)
MeSH Terms: conditions — Melanoma | interventions — Interferon-alpha

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Drug: recombinant interferon alfa

SUMMARY:
This randomized phase III trial is studying high dose interferon alfa to see how well it works compared to observation only in treating patients with stage II or stage III melanoma that has been completely removed by surgery.

DETAILED DESCRIPTION:
Interferon alfa may interfere with growth of cancer cells. It is not yet known whether treatment with interferon alfa is more effective than observation alone for stage II or stage III melanoma that has been completely removed surgically.

ELIGIBILITY:
Inclusion Criteria:

* Histologically confirmed primary melanoma of cutaneous origin
* Stage II (T3 N0 M0 1.5-4.0mm Breslow depth
* Clinically negative regional lymph node pathologic status unkown OR
* Histologically negative regional lymph nodes
* Stage III (T4 N0 M0)
* Greater than 4.0mm Breslow depth OR
* Stage III (T1-4 N1)
* One lymph node positive microscopically
* Patients must meet at least 1 of the following criteria
* T2b N0 primary melanoma 1.01-2.0mm with ulceration, node negative
* T3a-b N0 primary melanoma 2.01-4.0mm with and without ulceration, node negative
* T4a-b N0 primary melanoma > 4.0mm with and without ulceration, node negative
* T1aN1a-2a (microscopic)-primary melanoma of any thickness with microscopically positive lymph node (any number)
* Note EORTC patients who are node negative T2 or T3 are ineligible
* Patients with positive sentinel node should undergo complete lymphadenectomy of the nodal basin prior to study
* Must complete all primary therapy (wide excision with or without lymphadenectomy) and be randomized in the study within 84 days of wide excision
* No clinical, radiological/laboratory, or pathological evidence of incompletely resected melanoma or any distant metastatic disease
* No clinically palpable lymphadenopathy

Age:

* 18 and over

Performance Status:

* ECOG 0-1

Life expectancy:

* Not specified Hematopoietic
* WBC at least 3,000/mm^3
* Platelet count at least 125,000/mm^3
* Hematocrit at least 30%

Hepatic:

* Bilirubin no greater than 2 times the upper limit of normal (ULN)
* AST, LDH, and Alkaline phosphate no greater than 2 times ULN
* If lactate dehydrogenase or alkaline phosphate is above normal, a contrast enhanced CT scan or MRI of the liver is required to document the absence of tumor

Renal:

* BUN no greater than 33mg/dl OR
* Creatinine no greater than 1.8mg/dl

Cardiovascular:

* No history of active ischemic heart disease
* No cerebrovascular disease
* No congestive heart failure(New York Heart Association class III or IV heart disease)

Exclusion Criteria:

Biologic Therapy:

* No prior immunotherapy including tumor vaccines, interferon, interleukins,levamisole, or other biologic response modifers for melanoma Chemotherapy
* No prior or concurrent chemotherapy Endocrine Therapy
* No concurrent systemic corticosteriods including oral steriods (i.e., prednisone, dexamethasone), topical steroid creams or ointments, or any steriod-containing inhalers.

Radiotherapy:

* No Prior or concurrent radiotherapy

Surgery:

* See Disease characteristics

Other:

* No other concurrent immunosuppressive medications
* No other history of invasive melanoma
* No autoimmune disorders or conditions of immunosuppression
* No other concurrent or prior malignancies within past 5 years
* Cancer in situ
* Lobular carcinoma in situ of breast
* Carcinoma in situ of the cervix
* Atypical melanocytic hyperplasia or Clark 1 melanoma in situ
* Basal or squamous cell skin cancer
* No evidence of organic brain syndrome or significant impairment of basal cognitive function or any psychiatric disorder that would preclude study participation
* No other significant medical or surgical condition, or any medication or treatment regimens, that would interfere with study participation.
* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use effective contraception during and for 6 months after study

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2000-01

CONTACTS AND LOCATIONS:
Overall Officials: David S. Siegel, MD, Principal Investigator — Hackensack Meridian Health
Locations (1):
- The Cancer Center at Hackensack University Medical Center, Hackensack, New Jersey, United States

REFERENCES:
- [Derived] Slawek-Szmyt S, Araszkiewicz A, Jankiewicz S, Grygier M, Mularek-Kubzdela T, Lesiak M. Outcomes With Hybrid Catheter-Directed Therapy Compared With Aspiration Thrombectomy for Patients With Intermediate-High Risk Pulmonary Embolism. Cardiovasc Drugs Ther. 2025 Oct;39(5):1201-1213. doi: 10.1007/s10557-024-07562-4. Epub 2024 Apr 2. PMID 38564122